CLINICAL TRIAL: NCT05336370
Title: Decoding Mechanisms of Pain Modulation Through Hypnosis and Vagus Nerve Stimulation
Brief Title: Decoding Mechanisms of Pain Modulation
Acronym: HypnoPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Silje Endresen Reme, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 409472
Record Dates: First submitted 2022-04-12; First posted 2022-04-20 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain | interventions — Hypnosis; Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: The HypnoPain trial is designed as an experimental randomized controlled, statistician blinded superiority trial with three parallel groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The two vagus nerve stimulation arms are double-blinded, both for the participants and the outcome assessor, whilst the hypnosis arm is not possible to blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Hypnosis (Experimental): A brief hypnosis session will be provided to participants in this arm prior to immersion in the cold water.
  Interventions: Behavioral: Hypnosis
- Active tVNS (Experimental): Participants in the active tVNS condition will receive electronic stimulation of the vagus nerve prior to immersion in the cold water.
  Interventions: Device: Vagus nerve stimulation
- Sham tVNS (Sham Comparator): Participants in the sham tVNS will receive the electrode similar to the active treatment, but no stimulation will be performed.
  Interventions: Device: Sham control

INTERVENTIONS:
Behavioral: Hypnosis — The hypnosis will be conducted by clinical psychologists who have the formal competence and training in hypnosis. We will be using a tailored hypnosis script designed for this particular study, with a duration of 10-15 minutes. The script involves a hypnotic induction (relaxation-based), imagery (suggestions for pleasant visual imagery), a deepening procedure, and symptom-specific suggestions. The introduction begins by having the hypnotist debunk many of the common myths and misconceptions that patients may hold about hypnosis, and provide a description of hypnosis. Hypnosis is described as focused attention and concentration - like being so lost in a book or movie that it is easy to lose track of what is going on around you. Once the patient is deeply hypnotized, the therapist offers suggestions to reduce distress and improve pain tolerance.
  Arms: Hypnosis
Device: Vagus nerve stimulation — A CE approved tVNS device will be used to stimulate the afferent auricular branch of the vagus nerve located medial of the tragus at the entry of the acoustic meatus [36]. A standardized intensity of 10 mA with a pulse width of 250 μs and a consistent stimulation frequency of 25 Hz will be used for optimal stimulation. The stimulation will constantly alternate between active stimulation for 30 seconds, followed by a break of 30 seconds [37], and will have a duration of 15 minutes. Active tVNS is performed in a relaxed position, sitting back in a chair no more than 30 degrees from the horizontal, with both feet flat on the floor, and hands on thighs with palms facing downward. The bipolar stimulation electrode is placed correctly within the concha of the left ear. Participants are instructed to breathe normally while not talking or making any movements during their session.
  Arms: Active tVNS
Device: Sham control — Sham tVNS is performed in a relaxed position, sitting back in a chair no more than 30 degrees from the horizontal, with both feet flat on the floor, and hands on thighs with palms facing upward. The bipolar stimulation electrode is placed correctly within the concha of the left ear, but no actual stimulation will be performed. The electrode will be left on for 15 minutes. Participants are instructed to breathe normally while not talking or making any movements during their session
  Arms: Sham tVNS

SUMMARY:
The main objective of this experimental trial is to gain further insights into the mechanisms of pain modulation, and more specifically, whether expectations of coping is one of the involved mechanisms. This will be investigated by comparing two different interventions known to influence pain perception; hypnosis and non-invasive stimulation of the vagus nerve, prior to a pain exposure task (hand immersion in cold water). Expectations will be assessed both pre- and post intervention.

DETAILED DESCRIPTION:
Pain is a subjective experience, influenced by biological, psychological and social factors. This multidimensional view of pain has led to various efforts to affect people's pain experience. Nonpharmacological interventions, such as hypnosis, have proven successful in reducing pain whilst providing few, if any, negative side effects. Hypnosis involves a state of highly focused attention, with a constriction in peripheral awareness and a heightened responsiveness to social cues. This particular state can exert a powerful influence on the mind and body, yet the mechanisms responsible for this effect remains to a large degree unknown. The aim of this study is to investigate the effect of hypnosis given prior to a painful procedure (cold pressor test, CPT), to investigate the effect on pain perception and tolerance, but most importantly, to investigate if the effect is mediated by a change in expectations of coping. Previous studies have provided support for the the effect of hypnosis on expectations, but they have focused exclusively on stimulus expectancies (expectations of pain intensity), while the current study will focus on response outcome expectancies (expectations of coping) in line with the Cognitive Activation Theory of Stress (CATS).

Whilst hypnosis may dampen the stress response through expectancies (top-down), another way of dampening the stress response is through transcutaneous vagus nerve stimulation (tVNS) (bottom-up). Vagus nerve stimulation is proposed as another nonopioid pain treatment with minimal side effects. The vagus nerve is the 10th cranial nerve, connecting the viscera and the brain and influencing multiple systems of the body including the cardiac, immunologic, and endocrine system, and the activity of many visceral organs. This makes the vagus nerve a possibly important mediating (transmitting) and modulating nerve of pain signals . Stimulation of the vagus nerve is believed to modulate pain by inhibiting inflammation, oxidative stress, and sympathetic activity, and possibly also by inducing a brain activation pattern that may be incongruent with the pain matrix (i.e. brain regions commonly active during pain). VNS might also mediate the effects of the opioid system in pain modulation. These mechanisms have in common that they are hypothesized to affect neuronal hyperexcitability, resulting in a reduced pain perception, which is supported by experimental animal studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-70 years
* Fluent Norwegian language skills

Exclusion Criteria:

* History of cardiovascular disease
* Chronic pain conditions (any diagnoses resulting in chronic pain)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Pain tolerance | up to 10 minutes (During exposure (hand immersion in cold water))
  Time elapsed before removing the hand from the water.

SECONDARY OUTCOMES:
Pain intensity | Immediately after the cold pressor test
  rated on a NRS 0-10 where 0 is "no pain" and 10 is "the worst pain imaginable"
Pain bothersomeness | Immediately after the cold pressor test
  NRS 0-10 where 0 is "not bothersome at all" and 10 is "the most bothersome imaginable"

OTHER OUTCOMES:
Expectancies of coping | Within 5 minutes pre- and within 5 minutes post intervention
  NRS 0-10: "To what degree do you expect to cope with the painful procedure?"
Expectancies of coping: pre-conscious | Within 5 minutes pre- and within 5 minutes post intervention
  The Function Acquisition Speed Test, linking verbal associations involving the painful procedure (CPT) and coping concordant and dis-concordant words

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the study protocol, README files as well the statistical codes for the main analysis in an open repository (e.g. Open Science Framework) to ensure transparency and reproducability.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: As soon as possible
Access Criteria: Openly accessible

REFERENCES:
- See also: Related Info — https://www.uio.no/for-ansatte/arbeidsstotte/forskningsstotte/forskpro/prosjekter/sv/psi/Hypnose-og-vagusnervestimulering-for-smertetest/index.html